CLINICAL TRIAL: NCT06362837
Title: Realizing Gender Equality, Attitudinal Change & Transformative Systems in Nutrition (REACTS-IN)
Brief Title: Evaluation of REACTS-IN, an Intervention to Improve Nutrition, Hygiene, and Sexual and Reproductive Health Services
Acronym: REACTS-IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: World Vision Canada (Other); Global Affairs Canada (Other)
Responsible Party: Principal Investigator, Grace S. Marquis, Associate Professor, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P0117910-001
Record Dates: First submitted 2024-04-04; First posted 2024-04-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Stunting; Gender Equality; Acceptability of Health Care; Diet; Deficiency; Empowerment
Keywords: nutrition; gender equity; health services; sexual and reproductive rights; dietary diversity; anthropometry; sexual and reproductive health services; WASH
MeSH Terms: conditions — Growth Disorders; Patient Acceptance of Health Care; Malnutrition; Empowerment; Coitus | interventions — Gender Equity; Therapeutic Irrigation; Sex; Health

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental design for the evaluation of an intervention that is in the community (including schools) as well as in the local health service facilities. The data collection at baseline, midline, and end-line will occur simultaneously in the intervention and comparison selected communities. Comparison communities will not be visited during midline. Participants are unique at each time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Includes multiple activities, depending on country, including support of school-based iron-folic acid supplementation program; promotion of bio-fortified crops (sweet potatoes, beans, rice, corn); training on nutrition, water & sanitation, gender equity for rural communities through community groups and for health facility staff; support to improve gender-sensitive health services for nutrition, sexual and reproductive health,
  Interventions: Behavioral: Education intervention on nutrition, gender equity, WASH, sexual and reproductive health rights; Dietary Supplement: school-based iron-folic acid supplement program; Behavioral: Health service training on equitable access to nutrition, health, and sexual and reproductive services; Dietary Supplement: bio-fortified crops
- Comparison (No Intervention): No intervention will take place. Standard of care will be available in the health facilities and schools.

INTERVENTIONS:
Behavioral: Education intervention on nutrition, gender equity, WASH, sexual and reproductive health rights — Educational training on nutrition, gender equity, WASH, sexual and reproductive health rights will take place in communities (including schools) for women, men, and adolescents
  Arms: Intervention
Dietary Supplement: school-based iron-folic acid supplement program — The program will help support and promote the school-based programs of weekly iron and folic acid supplementation for adolescent girls, in countries where it is allowed.
  Arms: Intervention
Behavioral: Health service training on equitable access to nutrition, health, and sexual and reproductive services — Training and support activities to make gender-equitable nutrition, health, and sexual and reproductive services in the health facilities
  Arms: Intervention
Dietary Supplement: bio-fortified crops — The program promotes and distributes bio-fortified crops, including orange-fleshed sweet potatoes, rice, beans, and corn
  Arms: Intervention

SUMMARY:
This is an independent evaluation of World VIsion's 7-year quasi-experimental intervention to improve nutrition, nutrition-related rights and gender equality for women, adolescent girls, and children under five years of age in rural Bangladesh, Kenya, and Tanzania. The evaluation will collect baseline, midline, and end-line data from intervention communities, schools, and health facilities. Only baseline and endline will be collected on the comparison communities. The evaluation objectives are to test if the intervention improved indicators for (i) child anthropometry, (ii) maternal and child dietary practices, (iii) women's empowerment, and (iv) equitable health service access for nutrition and sexual and reproductive needs. The evaluation analysis will take into account gender differences in the indicators.

DETAILED DESCRIPTION:
This is an independent evaluation of World VIsion's 7-year quasi-experimental intervention ("Realizing Gender Equality, Attitudinal Change and Transformative Systems in Nutrition", REACTS-IN) to improve nutrition, nutrition-related rights and gender equality for women, adolescent girls, and children under five years of age in rural Bangladesh, Kenya, and Tanzania. REACTS-IN is a multi-sectoral approach, integrating nutrition-related determinants, such as water, sanitation, and hygiene (WASH) interventions and health systems strengthening, to improve access to quality and gender-responsive health systems with increased capacity to prevent and treat malnutrition, especially at the primary health care level. REACTS-IN includes both nutrition-specific (e.g., school-based iron-folic acid supplement program) and nutrition-sensitive (e.g., WASH education) activities delivered through local health systems and/or schools, and communities.

This independent evaluation will include three data collection at baseline, midpoint, and end-line to evaluate the performance indicators for the ultimate and intermediate outcomes. This includes indicators for child anthropometry, maternal and child dietary practices, women's empowerment, and equitable health service access for nutrition and sexual and reproductive needs. The evaluation analysis will take into account gender differences in the indicators.

The data collection will be carried out with intervention communities as well as with comparison communities. The estimated household sample is 463 households (women, husbands, child)/arm/country per time point, selected through a multi-stage cluster sampling methodology. The household baseline survey with a representative sample of mothers with children (0-5.9 mo; 6-23.9 mo; 24-59.9 mo) will be compared to the values at midpoint (to assess initial impact and the need for program adjustments) and at end-line (to assess the total impact of the project). The surveys will include sociodemographic, economic, and environmental information to assess the indicators for the local context. The evaluation also includes a sample of 500 school-going adolescents (250 boys, 250 girls)/arm/country per time point to assess indicators of knowledge about nutrition, menstrual hygiene management, and sexual and reproductive health. Finally, a sample of approximately 24 health staff and community leaders will provide qualitative data on gender-equitable access to services per arm/country for baseline and end-line.

Although the project also is working in Somalia, this independent evaluation does not include data collection in Somalia.

ELIGIBILITY:
Inclusion Criteria:

(i)Women:

* 15-49 y of age
* biological mother of child in the home who is 0-5.9, 6-23.9, or 24-59.9 months
* has lived in the community for at 12 months

(ii) Husbands/partners:

* no age limit
* lives in the home with index woman
* has lived in community for at least 12 months

(iii) Adolescents:

* 10-19 years
* male or female
* has been in target school for at least 6 months
* lives in the target community

(iv) Children:

* 0-5.9, 6-23.9, or 24-59.9 months

Exclusion Criteria:

(i) Children:

* no limitation on normal diet or growth (birth defects, illnesses)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13500 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-05-24 (Estimated)

PRIMARY OUTCOMES:
Gender equality | Change between baseline and study completion, an average of 5 years
  Percent of households with children < 59.9 mo that have achieved gender equality
Child anthropometry | Change between baseline and study completion, an average of 5 years
  Percent of children 6-59 mo of age who are stunted

SECONDARY OUTCOMES:
Antenatal care | Change between baseline and study completion, an average of 5 years
  Percent of mothers of children 0-6 months who attended at least four ante-natal visits during the last pregnancy from skilled health personnel
Contraception use by women and partners | Change between baseline and study completion, an average of 5 years
  Percent of women aged 15-49 years married or in union, who are currently using, or whose sexual partner is using at least one modern contraception method
Child diet | Change between baseline and study completion, an average of 5 years
  Percent of children 6-23.9 months of age, who receive minimum dietary diversity and minimum meal frequency
Sexual and reproductive health services for adolescents | Change between baseline and study completion, an average of 5 years
  Percent of adolescent girls (10-19) who report that they were offered sexual and reproductive health services
Gender equitable health services for nutrition, health, and sexual and reproductive health | Change between baseline and study completion, an average of 5 years
  Percent of health facilities promoting gender equitable and responsive nutrition, health, and sexual and reproductive services
Exclusive breastfeeding | Change between baseline and study completion, an average of 5 years
  Percent of children 0-5.9 mo who are exclusively breastfed
Use of family planning | Change between baseline and study completion, an average of 5 years
  Percent of women 15-49 y who decided to use family planning
adolescent knowledge of nutrition, menstrual hygiene, and sexual and reproductive health | Change between baseline and study completion, an average of 5 years
  Percent of adolescent girls and boys with appropriate knowledge about nutrition, menstrual hygiene, and sexual and reproductive health
maternal knowledge on nutrition | Change between baseline and study completion, an average of 5 years
  Percent of women 15-49 y with appropriate knowledge on good maternal nutrition
Attended birth deliveries | Change between baseline and study completion, an average of 5 years
  Percent of deliveries attended by skilled birth personnel
maternal knowledge of family planning | Change between baseline and study completion, an average of 5 years
  Percent of mothers who know at least 3 modern methods of family planning
maternal knowledge of exclusive breastfeeding | Change between baseline and study completion, an average of 5 years
  Percent of mothers who know at least 3 benefits of exclusive breastfeeding
mothers planting biofortified crops | Change between baseline and study completion, an average of 5 years
  Percent of mothers who have planted biofortified crops from REACTS-IN materials
mothers planting nutrient dense local vegetables | Change between baseline and study completion, an average of 5 years
  Percent of mothers who have planted nutrient dense local vegetables from REACTS-IN seeds
mothers planting trees | Change between baseline and study completion, an average of 5 years
  Percent of mothers who have planted fruit tress from REACTS-IN materials
hygenic toilets | Change between baseline and study completion, an average of 5 years
  Percent of households with hygienic toilets
community health worker visit | Change between baseline and study completion, an average of 5 years
  Percent of households that received at least one community health worker visit in last month
Adolescent iron folic acid supplements | Change between baseline and study completion, an average of 5 years
  Percent of adolescent girls who received the recommended scheme of weekly iron-folic actic supplements
health facility | Change between baseline and study completion, an average of 5 years
  Percent of health facilities scoring > 80 on planning assessment

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Marquis, PhD, Principal Investigator — McGill University
Locations (3):
- Brac University, Dhaka, Bangladesh
- Connar Consultants, Nairobi, Kenya
- Ifakara Health Institute, Ifakara, Tanzania

IPD SHARING:
Plan to Share IPD: No